CLINICAL TRIAL: NCT05751902
Title: Translation and Validation of the Arabic Version of the Oral Health Impact Profile Questionnaire
Brief Title: Translation and Validation of the Arabic Version of the OHIP Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Medhat Sameh Abdelaziz, Assistant Lecturer of Prosthodontics, Future University in Egypt
Other Study IDs: FUE.REC (1)/1-2023
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Oral Health; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Arabic version of OHIP questionnaire — Translated Arabic version of Oral Health Impact Profile questionnaire

SUMMARY:
OHIP questionnaire was originally developed in English and in order to make use of this tool to measure the oral health-related quality of life of elderly Arabic populations, A translation is necessary. Also, validation of the translated instrument is very important. As people living in middle east are mainly influenced by the Arabic culture, which differs significantly from the Western culture where the OHIP questionnaire was first developed.

254 participants having removable prosthesis will be asked to complete translated Arabic version of OHIP questionnaire for validation.

ELIGIBILITY:
Inclusion Criteria:

* Patients having removable partial denture in the last year
* Native Arabic patients

Exclusion Criteria:

* Patients non familiar with Arabic language
* patients with mental or perception problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: any participant fluent in Arabic language and having a removable prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-01-28 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Reliability and validity | 3 months
  Reliability of Translated Arabic version of OHIP questionnaire using internal consistency

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided